CLINICAL TRIAL: NCT02196155
Title: Botulinum Toxin A Versus Steroids for the Treatment of Chronic Plantar Fasciitis: a Randomized Controlled Study
Brief Title: Botulinum Toxin A Versus Steroids for the Treatment of Chronic Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32003B_152671
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; Botulinum toxin A; Cortisone; RCT
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Botulinum Toxins, Type A; Cortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BTX-A (Active Comparator): Botulinum A toxin is injected each 100 U in both gastrocnemius muscle-bellies and 50 U in the soleus muscle, i.e. a total of 250 U.
  Interventions: Drug: Botulinum toxin A
- Cortisone (Active Comparator): Depot Medrol is injected at the plantar fascia insertion site at the calcaneus
  Interventions: Drug: cortisone
- Saline (Placebo Comparator): Placebo saline is injected in both gastrocnemius muscle-bellies and in the soleus muscle
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum toxin A — Researchers discovered in the 1950s that injecting overactive muscles with minute quantities of botulinum toxin type-A would result in decreased muscle activity. Botulinum toxin type-A has this effect because it prevents the vesicle where the acetylcholine is stored from binding to the membrane where the neurotransmitter can be released. Botulinum toxin type-A thus blocks the release of acetylcholine by the neuron. This will effectively weaken the muscle for a period of three to four months.
  In addition to its cosmetic applications, Botox is currently used in the treatment of spasms and dystonias, by weakening involved muscles, for the 60-70 day effective period of the drug. The main conditions treated with botulinum toxin are: Cervical dystonia (spasmodic torticollis) (a neuromuscular disorder involving the head and neck), Blepharospasm (excessive blinking) etc..
  Arms: BTX-A
Drug: cortisone
  Arms: Cortisone
Drug: Saline
  Arms: Saline

SUMMARY:
Plantar fasciitis is the classic and most common type of heel pain. Considering the costs for health care and the temporary disability not only for work, plantar fasciitis results in a substantial (and at least partially unnecessary) burden for the Swiss health care system and national economics.

Nonoperative treatment is the mainstay of treating plantar fasciitis. However, so far no treatment has proven to be superior to others, and there is national and international lack of consensus of how to treat plantar fasciitis best.

The investigators believe that the BTX-A injection in the gastrocnemius and the soleus muscles is currently the most promising non-operative approach, because it is considered to treat the disease at its origin (temporary weakening of the tight triceps surae muscle) as opposed to simply alleviate the symptoms (e.g. plantar cortisone and other injections, ESWT).

However, to date there is no evidence in the literature that compares the new, promising technique of BTX-A injection into the gastroc-soleus complex to a sham (saline) injection and to the gold standard steroid injection at the plantar fascia insertion site. With the intended study, this gap is going to be closed.

DETAILED DESCRIPTION:
Background

Plantar fasciitis is the classic and most common type of heel pain. Extrapolating the rate of 2 million or 0.6% of the US American population being treated for plantar fasciitis every year to Switzerland, the corresponding number of patients would amount to 50'000 patients being treated for plantar fasciitis. Considering the costs for health care and the temporary disability not only for work, plantar fasciitis results in a substantial (and at least partially unnecessary) burden for the Swiss health care system and national economics.

Nonoperative treatment is the mainstay of treating plantar fasciitis. In the literature, numerous operative and nonoperative treatment approaches for plantar fasciitis have been suggested. However, so far no treatment has proven to be superior to others, and there is national and international lack of consensus of how to treat plantar fasciitis best. Numerous prescriptions for unnecessary orthoses, expensive and painful shock waves, and complications following steroid injection could be obviated, when the safe BTX-A injection demonstrates good results.

The investigators believe that the BTX-A injection in the gastrocnemius and the soleus muscles is currently the most promising non-operative approach, because it is considered to treat the disease at its origin (temporary weakening of the tight triceps surae muscle) as opposed to simply alleviate the symptoms (e.g. plantar cortisone and other injections, ESWT).

The high number of level I and II studies suggests that there is need for clarification and evaluation of the efficacy of several non-operative and operative treatment approaches for the chronic plantar fasciitis. However, to date there is no evidence in the literature that compares the new, promising technique of BTX-A injection into the gastroc-soleus complex to a sham (saline) injection and to the gold standard steroid injection at the plantar fascia insertion site. With the intended study, this gap is going to be closed. Objective evaluation of the BTX-A efficacy includes the randomized allocation of patients to the BTX-A, the steroid, or the saline group, the blinded comparison to the sham (saline) injection, and finally the MRI assessment at the beginning and at the end of the followup. With the evidence resulting from this study, patients can be superiorly counseled in the future with regard to efficacy of nonoperative treatment of plantar fasciitis.

Objective

Plantar fasciitis is the classic and most common type of heel pain. Considering the costs for health care and the temporary disability not only for work, plantar fasciitis results in a substantial (and at least partially unnecessary) burden for the Swiss health care system and national economics. However, so far no treatment has proven to be superior to others, and there is national and international lack of consensus of how to treat plantar fasciitis best.

Methods

Patients are randomly allocated to three groups (1 - 3).

- Patient group 1 - combination of physiotherapy, stretching exercises according to DiGiovanni et al and BTX-A injection into the gastroc-soleus complex: One hundred units (U) of toxin are applied to each muscle belly, and 1 application of 50 U is administered to the soleus, making a total of 250 U.

* Patient group 2 - physiotherapy, stretching exercises according to DiGiovanni combined with cortisone injection into the plantar fascia
* Patient group 3 - physiotherapy, stretching exercises according to DiGiovanni and saline injection into the gastroc-soleus complex (sham control group)

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of a plantar fasciitis
* Plantar fasciitis in MRI
* Exclusion of differential diagnoses
* Symptoms more than 3 months
* Absolution of 3 months unsuccessful treatment
* Written informed consent

Exclusion Criteria

* Active differential diagnoses
* Contraindications: pregnancy and breastfeeding, infection at injection sites, allergy against BTX-A
* Previous injections or surgery for plantar fasciitis
* Neurological diseases affecting the peripheral nervous system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in foot pain | at 6 weeks, 3, 6 and 12 (24) months
  Measured by VAS FA subjective foot score

SECONDARY OUTCOMES:
Change from baseline in patient health | at 6 weeks, 3, 6 and 12 (24) months
  Measured by SF 36
Change from baseline in pain, disability and activity restriction in foot | at 6 weeks, 3, 6 and 12 (24) months
  Measured by foot functional index FFI
General pain | at 6 weeks, 3, 6 and 12 (24) months
  Measured by VAS pain scale
Reduction of inflammation | pre-intervention and at 12 months
  Measured by MRI
Number of patients with complications | at 6 weeks, 3, 6 and 12 (24) months
Change from baseline in ankle range of motion | at 6 weeks, 3, 6 and 12 (24) months
  Measured by goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Krause, PD Dr., Principal Investigator — Dep. of Orthopaedic Surgery, Inselspital, University of Berne, Freiburgstrasse, 3010 Berne, Switzerland
Locations (2):
- Switzerland (2):
  - Dep, of Orthopaedic Surgery, Inselspital, University of Berne, Bern
  - Department of Orthopaedic Surgery, Kantonsspital Lucerne, Lucerne

REFERENCES:
- [Result] Brin MF, Lew MF, Adler CH, Comella CL, Factor SA, Jankovic J, O'Brien C, Murray JJ, Wallace JD, Willmer-Hulme A, Koller M. Safety and efficacy of NeuroBloc (botulinum toxin type B) in type A-resistant cervical dystonia. Neurology. 1999 Oct 22;53(7):1431-8. doi: 10.1212/wnl.53.7.1431. PMID 10534247
- [Result] Bihari K. Safety, effectiveness, and duration of effect of BOTOX after switching from Dysport for blepharospasm, cervical dystonia, and hemifacial spasm dystonia, and hemifacial spasm. Curr Med Res Opin. 2005 Mar;21(3):433-8. doi: 10.1185/030079905X36396. PMID 15811212
- [Result] Elizondo-Rodriguez J, Araujo-Lopez Y, Moreno-Gonzalez JA, Cardenas-Estrada E, Mendoza-Lemus O, Acosta-Olivo C. A comparison of botulinum toxin a and intralesional steroids for the treatment of plantar fasciitis: a randomized, double-blinded study. Foot Ankle Int. 2013 Jan;34(1):8-14. doi: 10.1177/1071100712460215. PMID 23386757